CLINICAL TRIAL: NCT06081478
Title: CD19/CD22 Bispecific CAR-T Cell Therapy for Relapsed/Refractory B-cell Lymphoma or Acute Lymphoblastic Leukemia: a Prospective, Single-arm, Single-center, Phase 2 Clinical Trial
Brief Title: CD19/CD22 Bispecific CAR-T Cell Therapy for Relapsed/Refractory B-cell Lymphoma or Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, LIANG WANG, Director of the department of hematology, Beijing Tongren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T001/TR
Record Dates: First submitted 2023-10-07; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; B-cell Lymphoma; Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19/CD22 CAR-T group (Experimental): Patients would receive autologous CAR-T cell therapy targeting both CD19 and CD22. The dosage for CD19-CAR-T cell was 2×10e6/kg and CD22-CAR-T cell was 1×10e6/kg. Both CAR-T cells were infused at the same day.
  Interventions: Drug: CD19/CD22-bispecific CAR-T cells

INTERVENTIONS:
Drug: CD19/CD22-bispecific CAR-T cells — CD19/CD22-bispecific CAR-T cells were infused at the same day with 2×10e6/kg and 1×10e6/kg dosage, respectively.

SUMMARY:
CAR-T cell therapy targeting CD19 has been shown to be effective in heavily-pretreated B-cell ALL or NHL, but relapses post-CAR-T are common, and CD19 antigen loss is one of the reasons. Thus, we supposed that CD19/CD22 bispecific CAR-T cell therapy would be more effective and less relapses would occur in B-ALL or NHL. In this prospective phase 2 clinical trial, we aim to explore the efficacy and safety of CD19/CD22 bispecific CAR-T cell therapy in relapsed/refractory B-ALL or Large B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 14 years to 85 years, expected survival > 3 months;
* CD19/CD22 positive B-cell lymphoma or B-ALL;
* relapsed or refractory to standard first-line treatment;
* ECOG-PS score=0-2;
* Having at least one measurable lesions;
* Cardiac function: 1-2 levels;
* Liver: TBIL≤3ULN，AST ≤2.5ULN，ALT ≤2.5ULN;
* kidney: Cr≤1.25ULN;
* bone marrow: WBC ≥ 3.0×10e9/L, Hb ≥80 g/L, PLT ≥ 50×10e9/L;
* No serious allergic constitution;
* No other serious diseases that conflicts with the clinical program;
* No other cancer history;
* No serious mental disorder;
* Informed consent is signed by a subject or his lineal relation.

Exclusion Criteria:

* Pregnant or lactating women; (female participants of reproductive potential must have a negative serum or urine pregnancy test);
* Uncontrolled active infection, HIV infection, syphilis serology reaction positive;
* Active hepatitis B or hepatitis C infection;
* Recent or current use of glucocorticoid or other immunosuppressor;
* With severe cardiac, liver, renal insufficiency, diabetes and other diseases;
* Participate in other clinical research in the past three months;
* previously treatment with any gene therapy products;
* Researchers think of that does not fit to participate in the study, or other cases that affect the clinical trial results.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Best ORR | From the day of CAR-T cells infusion to 3 months post-CAR-T cells infusion
  Overall response rate means sum of complete response rate and partial response rate

SECONDARY OUTCOMES:
Best CR rate | From the day of CAR-T cells infusion to 3 months post-CAR-T cells infusion
  CR was defined as complete remission evaluated using PET-CT scan or BM test
Progression free survival (PFS) | From the day of CAR-T cells infusion to 12 months post-CAR-T cells infusion
  PFS was defined from the date of CAR-T infusion to the date fo confirmed disease progression or death of any reason
overall survival (OS) | From the day of CAR-T cells infusion to 12 months post-CAR-T cells infusion
  OS was defined from the date of CAR-T infusion to the date fo death

CONTACTS AND LOCATIONS:
Locations (1):
- Liang Wang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No